CLINICAL TRIAL: NCT01726530
Title: Transdermal Fentanyl Patch for Postoperative Analgesia After Abdominal Surgery: a Randomized Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE541094
Record Dates: First submitted 2012-11-10; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Postoperative Pain Relief
Keywords: transdermal fentanyl patch, postoperative pain,
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdermal fentanyl patch (Active Comparator): Transdermal fentanyl patch, 50 mcg/hour, was attached to the patient's chest wall at 10 pm the day before surgery
  Interventions: Drug: transdermal fentanyl patch (50 mcg/hour)
- Placebo (Placebo Comparator): Placebo patch was attached to the patient's chest wall at 10 pm the day before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: transdermal fentanyl patch (50 mcg/hour)
  Other Names: Duragesic
  Arms: Transdermal fentanyl patch
Drug: Placebo
  Arms: Placebo

SUMMARY:
Abdominal surgery causes severe postoperative pain. Multi-modal pain therapy is usually applied but there is no perfect choice. It depends on physician's skill and situation. The best regimen is patient-controlled analgesia, but it requires an expensive equipment. Transdermal fentanyl patch, usually used in chronic pain relief, can steadily release fentanyl into blood stream for 72 hours, but it has slow onset of 12 hours.

Hypothesis: If Transdermal fentanyl patch is applied 10-12 hours before surgery, it may provide good analgesia for 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* age =>18 years
* scheduled for abdominal surgery

Exclusion Criteria:

* ASA class > 3
* Known allergy to fentanyl or morphine
* History of substance or alcohol abuse, and tolerance or dependence on opioids
* Combined epidural block
* Can't use PCA, abnormal renal / liver function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  Compare the cumulative morphine consumption during 24 hours postoperative of both study and control groups.

SECONDARY OUTCOMES:
morphine consumption | 48 and 72 hours
  Compare the cumulative morphine consumption during 48 and 72 hours postoperative of both study and control groups.

OTHER OUTCOMES:
side effects | 72 hours
  Compare the side effects, i.e.nausea, vomiting, itching, respiratory depression during 72 hours postoperative of both study and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD., Study Chair — Khon Kaen University
Locations (1):
- Srinagarind hospital, Khon Kaen, Changwat Khon Kaen, Thailand